CLINICAL TRIAL: NCT02069145
Title: A Phase 1b Dose Escalation Study of OMP-54F28 in Combination With Sorafenib in Patients With Hepatocellular Cancer
Brief Title: Dose Escalation Study of OMP-54F28 in Combination With Sorafenib in Patients With Hepatocellular Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54F28-004
Record Dates: First submitted 2014-02-18; First posted 2014-02-24 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Hepatocellular Cancer; Liver Cancer
Keywords: Hepatocellular Cancer; Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — OMP-54F28; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug: OMP-54F28, with Sorafenib (Experimental)
  Interventions: Drug: OMP-54F28 with Sorafenib

INTERVENTIONS:
Drug: OMP-54F28 with Sorafenib
  Other Names: OMP-54F28; Sorafenib

SUMMARY:
This is an open-label Phase 1b dose-escalation study to assess the safety, tolerability, and PK of OMP-54F28 when combined with sorafenib. OMP-54F28 will be administered IV on Day 1 of each 21-day cycle. The planned dose levels of OMP-54F28 are 5 and 10 mg/kg. Depending on safety in this study, additional lower or intermediate dose levels may be evaluated.

DETAILED DESCRIPTION:
Depending on emerging safety data from the Phase 1a study 54F28-001 with continuing dose escalation, additional higher dose levels of OMP-54F28 may be evaluated in this study. Alternative dosing schedules of OMP-54F28 may be explored based on emerging nonclinical and clinical data for safety, PD, PK and efficacy. The starting dose for a new dosing schedule will be chosen to result in an AUC equivalent to the highest dose level that cleared on the previously studied dosing schedule. No dose escalation of OMP-54F28 will be allowed within a dose cohort. Sorafenib 400 mg will be given orally twice daily (PO BID). Sorafenib dosing schedules with a total daily dose <800 mg (e.g. Sorafenib 400 mg once daily) may be evaluated in this study depending on emerging safety data from this study.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥18 years
* Histologically documented hepatocellular carcinoma
* Locally advanced or metastatic disease
* Availability of FFPE tumor tissue, either archival or obtained at study entry through fresh biopsy

  o Tumor tissue from fine needle aspiration is not acceptable.
* ECOG performance status of 0 or 1 (see Appendix C)
* All acute treatment-related toxicity from prior therapy must have resolved to Grade ≤ 1 prior to study entry
* Adequate hematologic and end-organ function
* Child-Pugh Classification A (see Appendix D)
* Evaluable or measurable disease per RECIST v1.1
* For women of childbearing potential and men with partners of childbearing potential, agreement to use two effective forms of contraception

Exclusion Criteria:

* Inability to take oral medications
* Prior systemic therapy for locally advanced or metastatic hepatocellular cancer
* Prior adjuvant therapy with sorafenib or another Raf/VEGF inhibitor
* Prior history of allografts, including, but not limited to, liver and bone marrow transplants
* Esophageal or gastric variceal bleeding within last 3 months
* Risk for varices, based on known history of esophageal or gastric varices, evidence of hepatic cirrhosis and/or portal hypertension including biopsy-proven cirrhosis, hypersplenism, or radiographic findings of varices
* Clinically evident ascites
* Evidence of encephalopathy within last 3 months
* Treatment with inducers of cytochrome P450 3A4 (CYP3A4) within 7 days prior to first dose of study treatment
* Treatment with interferon within 4 weeks prior to first dose of study treatment
* Treatment with any anti-cancer therapy, including radiotherapy, chemotherapy, biologic therapy, or herbal therapy within 3 weeks or 5 half-lives (for systemic agents), whichever is shorter
* Known hypersensitivity to any component of study treatments that resulted in drug discontinuation
* Uncontrolled seizure disorder or active neurologic disease
* Untreated brain metastases
* Leptomeningeal disease as a manifestation of cancer
* Active infection requiring antibiotics
* Bisphosphonate therapy for symptomatic hypercalcemia
* Significant intercurrent illness including, but not limited to, unstable angina pectoris, and cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements
* Pregnancy, lactation, or breastfeeding
* Known HIV infection
* Active Hepatitis B infection in the absence of adequate antiviral therapy
* Uncontrolled hypertension, defined as systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg, despite medical management
* Pulmonary hemorrhage of Grade ≥2 within 28 days prior to first dose of study treatment
* Any other hemorrhage or bleeding of Grade ≥3 within 28 days prior to first dose of study treatment
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Concurrent use of therapeutic warfarin
* New York Heart Association Classification III or IV (see Appendix F)
* Congenital long QT syndrome
* Known clinically significant gastrointestinal disease including, but not limited to, inflammatory bowel disease
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to the first dose of study treatment or anticipation of need for major surgical procedure during the course of the study
* Osteoporosis based on a T-score of <-2.5 at the left or right total hip, left or right femoral neck or lumbar spine (L1-L4) as determined by DEXA scan
* Bone metastases and one of the following:

  * Prior history of a pathologic fracture
  * Lytic lesion requiring an impending orthopedic intervention
  * Lack of treatment with a bisphosphonate or denosumab
* Treatment with a thiazolidinedione PPAR gamma inhibitor; e.g. Actos® (pioglitazone) and Avandia® (rosiglitzone)
* Active treatment with an oral or IV glucocortocoid for ≥4 weeks at a daily dose equivalent to or greater than 7.5 mg of oral prednisone
* Fasting β-CTX of >1000 pg/mL
* Metabolic bone disease, such as hyperparathyroidism, Paget's disease or osteomalacia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of OMP-54F28 in combination with sorafenib in patients with hepatocellular cancer | Subjects will be treated and observed for DLT through the end of the first cycle (from Day 0 - 21)
  The maximum tolerated dose (MTD) will be determined in patients treated with OMP-54F28 in combination with sorafenib in patients with hepatocellular cancer

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of OMP-54F28 and sorafenib when administered in combination to patients with hepatocellular cancer | OMP-54F28 will be administered IV on Day 1 of each 21 day cycle. Plasma sample for Parmacokinetics (PK) analysis to be obtained at various time points, 30 minutes after end of OMP-54F28 infusion and before sorafenib treatment
  Apparent half life, AUC, clearance, volume of distribution

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Massachussetts General Hospital, Boston, Massachusetts
  - Mount Sinai Medical Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania